CLINICAL TRIAL: NCT03235518
Title: A Combination HIV Prevention Strategy for Young Women at Risk for HIV
Acronym: IPrEP
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAAR0256; R01MH110051 (NIH)
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV Prevention; Female sex workers
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Structure Interviews with FSW: Structured interviews with 200 purposively sampled FSW will be conducted. These interviews will be conducted prior to focus group discussion (FGD) and in-depth qualitative interview (IDI) with FSW. Structured interviews will take approximately 45-60 minutes to complete and will be administered privately in Kiswahili, Dholuo or English by trained female research staff. Quantitative interviews will be administered to conduct an assessment of FSW sociodemographics, sexual behaviour patterns and HIV-related knowledge, attitudes and practices regarding HIV prevention and other factors that might affect initiation and adherence to PrEP use, ability to use PrEP covertly, HIV testing history, mobility patterns, social networks, pregnancy intentions, ability to use condoms consistently with clients, and regular partners, and interpersonal violence from clients, regular partners and the police.
- Focus Group Discussions with FSW: Three to five FGDs of up to 10 FSW per group will be conducted. These FGD will take place prior to FSW IDI. FSW who participated in FGDs will be ineligible for participation in the IDI. All group discussions will last approximately 1.5 to 2 hours and be conducted in Kiswahili, Dholuo or English. Each group discussion will be facilitated by trained female research staff and held in a private space at a pre-specified location. The themes that will be explored in the FGDs include: FSW social networks, participation in PrEP studies, barriers and facilitators to PrEP use and use of resource transfers for PrEP adherence. In addition, participants will complete a brief demographic survey.
- In-Depth Qualitative Interviews with FSW: 30 IDI will be conducted with FSW. FSW who participated in FGDs will be ineligible for participation in the IDI. All in-depth interviews will be conducted by trained female research staff using a semi-structured interview guide. All interviews will be held in a private space at a pre-specified location within the community. The topics that will be discussed in the IDI with FSW include demographics, social support, dynamics of sex work, HIV prevention methods (including condom use), perception of HIV risk and development of PrEP intervention.
- In-Depth Qualitative Interviews with MC: 30 IDI will be conducted with MC. All IDI will last approximately 60-90 minutes and be conducted in Kiswahili, Dholuo, or English. Each interview will be conducted by a trained male research staff using semi-structured interview guide. All interviews will be held in a private space at a pre-specified location. Topics include demographics, relationships with FSW, HIV prevention methods (including use of condoms), perception of HIV risk and development of PrEP intervention.
- In-Depth Qualitative Interviews with HCPs: 30 IDI will be conducted with health care provider (HCP). All IDI will last approximately 60-90 minutes and be conducted in English. Each interview will be conducted by trained research staff using a semi-structured interview guide. Interviews will be held in a private space at the health facility where they work or another venue preferred by the HCP. Topics include demographics, health care needs of FSW and sources of care, HIV prevention needs of FSW, PrEP for FSW and training needs for HCP.

SUMMARY:
The purpose of this study is to conduct formative research to inform the design and implementation of combination prevention interventions, including pre-exposure prophylaxis (PrEP) for female sex workers (FSW), as well as to inform recruitment and retention strategies for female sex workers and their male clients in Kenya.

DETAILED DESCRIPTION:
Despite remarkable advances in the global HIV response with 17 million persons, out of nearly 37 million living with HIV, who have initiated antiretroviral therapy (ART) in low- and middle-income countries (LMIC) as of end of 2015, there were an estimated 5,700 new HIV infections each day and a total of 2.1 million new HIV infections in 2015, of which 66% were in sub-Saharan Africa (SSA). Key populations within the generalized HIV epidemics in SSA, including female sex workers (FSW), have received insufficient attention, with data indicating that they are at disproportionate risk with limited access to prevention and treatment services. Globally, new infections among key populations and their sexual partners accounted for 36% of all new HIV infections in 2015. HIV prevalence among FSW is 29.3% worldwide. While reliable HIV prevalence estimates are lacking, younger FSW <25 years may be at significantly greater risk due to the confluence of biological, behavioral and structural risk factors.6 Mathematical modeling suggests that the proportion of new HIV infections attributable to sex work is likely to increase over time.

In settings where key populations contribute substantially to HIV burden, as in Kenya, effective integrated prevention strategies are urgently needed for populations such as FSW and can have a substantial impact on reducing new HIV infections.

In 2012, HIV prevalence among Kenyan 15-64 year olds was 5.6%, with 1,192,000 people living with HIV, but was markedly higher (15.1%) in the region of Kenya, formerly named Nyanza Province. HIV prevalence is 14.1% among FSW and 7.6% among male clients of sex workers (MC). FSW contribute significantly to new HIV infections in Kenya,14 with modelled estimates showing that 1 in 3 new HIV infections can be attributed to key populations.

ELIGIBILITY:
Inclusion Criteria:

FSW. Inclusion criteria for the structured interviews, FGDs and IDI are identical.

* Report being female or transgender women born make who have sex with men
* Report being HIV-negative or unknown status
* Report being between 18-24 years of age
* Report residing or working in study community
* Reports exchange sex for goods, money, flavors or other services in past 3 months
* Willing to allow audio-recording of FGDs or IDI
* Able to complete study procedures in English, Kiswahili or Dhuluo

Male Clients

* Male
* Report being >=18 years of age
* Report exchanging goods, money, favors or other services for sex in past 3 months
* Willing to allow audio-recording of IDI
* Able to complete study procedures in English, Kiswahili or Dhuluo

Health Care Providers

* Currently working as nurse or clinical officer at a clinic or other facility likely to offer PrEP
* Report being >= 18 years of age
* Willing to allow audio-recording of IDI
* Able to complete study procedures in English

Exclusion Criteria:

* Individuals who do not meet the inclusion criteria
* Individuals who in the opinion of the investigators would interfere with adherence to study study requirements
* FSW participating in FGD are not eligible for participation in IDI

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Female sex workers, male clients of female sex workers, and health care providers will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Percentage of FSW participants who would be willing to participate in HIV prevention research | 6 months
  To inform prevention interventions for FSW, we will assess the percentage of FSW willing to participate in HIV prevention research or a PrEP study

SECONDARY OUTCOMES:
Percentage of MC participants who would be willing to participate in HIV prevention research | 6 months
  To inform prevention interventions, we will assess the percentage of MC willing to participate in HIV prevention research

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa M. El-Sadr, MD, MPH, MPA, Principal Investigator — Columbia University
Locations (1):
- Kisumu, Kenya, Kisumu, Kenya